CLINICAL TRIAL: NCT05255965
Title: IL-8+ naïve T Cells as a Biomarker for Thymoma Identification: A Prospective, Multi-center Diagnostic Accuracy Study
Brief Title: IL-8+ naïve T Cells as a Biomarker for Thymoma Identification
Status: Completed | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-812
Record Dates: First submitted 2022-02-12; First posted 2022-02-25 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-02

CONDITIONS: Thymoma
Keywords: thymoma
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5ml peripheral venous blood was taken before surgery or biopsy, and the levels of initial T cell with IL-8+, PLXND1+, PTK7+ or CR2+ were detected and recorded within 6 hours, respectively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: level of IL-8+ initial T cells — 5ml peripheral venous blood was taken before surgery or biopsy, and the levels of initial T cell with IL-8+, PLXND1+, PTK7+ or CR2+ were detected and recorded within 6 hours, respectively.
  Other Names: level of PLXND1+ initial T cells; level of PTK7+ initial T cells; level of CR2+ initial T cells

SUMMARY:
According to the existing literature reports, the misdiagnosis rate of CT is as high as 22% - 68%. Thymic cyst and lymphoma are usually misdiagnosed as thymoma, resulting in many unnecessary operations; In addition, traditional imaging technologies can also cause a missed diagnosis rate of about 7%, which is common in the missed diagnosis of asymptomatic thymoma, which delays the opportunity of treatment. Therefore, in order to accurately treat thymic tumors, the existing diagnostic methods of thymic tumors need to be further optimized.

Our previous retrospective study found that the level of IL-8 + initial T cells can well distinguish thymoma from other types of anterior mediastinal tumors, and the sensitivity and specificity are close to 95%.

DETAILED DESCRIPTION:
This study is a prospective, multicenter diagnostic accuracy study. 310 patients with anterior mediastinal space occupying lesions who meet the enrollment conditions are planned to be recruited continuously. 5ml peripheral venous blood of the patients is taken before surgery or puncture biopsy and sent to the laboratory for blind detection of IL-8 + initial T cell level; Then the patient underwent anterior mediastinal tumor surgery or biopsy to obtain pathological results (gold standard for diagnosis). After the pathological results were confirmed, all cases were divided into thymoma group and non thymoma group. The sensitivity and specificity of IL-8 + initial T cells in the diagnosis of thymoma and the cutoff value of thymoma were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Adult, aged 18 and above；
* Patients with anterior mediastinal mass on imaging (chest CT or MRI)；
* The patient's anterior mediastinal mass can be diagnosed by biopsy or surgery.

Exclusion Criteria:

* Adolescents and children under the age of 18;
* The patient's anterior mediastinal mass can not be diagnosed by biopsy or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients who are clinically diagnosed with thymic masses.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
The sensitivity of levels of IL-8+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The specificity of levels of IL-8+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The cutoff value of levels of IL-8+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year

SECONDARY OUTCOMES:
The sensitivity of levels of PLXND1+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The specificity of levels of PLXND1+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The sensitivity of levels of PTK7+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The specificity of levels of PTK7+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The sensitivity of levels of CR2+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The specificity of levels of CR2+ initial T cells in the diagnosis of thymoma | Through study completion, an average of 2 year
The sensitivity of enhanced CT/MRI in the diagnosis of thymoma | Through study completion, an average of 2 year
The specificity of enhanced CT/MRI in the diagnosis of thymoma | Through study completion, an average of 2 year
The sensitivity of levels of IL-8+, PLXND1+, PTK7+ and/or CR2+ initial T cells combined with enhanced CT/MRI in the diagnosis of thymoma | Through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Jianyong Ding, Study Chair — Zhongshan Hospital Attached To Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: No